CLINICAL TRIAL: NCT01844362
Title: Prospective Case Series of Human Uterus Transplantation From Live Donor
Brief Title: Uterus Transplantation From Live Donor
Acronym: utx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Mats Brännström, Professor, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: utx-ld
Record Dates: First submitted 2013-04-23; First posted 2013-05-01 (Estimated); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Primary Uterine Infertility
Keywords: uterus; transplantation; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Uterine transplantation (Experimental): Patients undergo transplantation of the uterus from live donor.
  Interventions: Procedure: uterine transplantation

INTERVENTIONS:
Procedure: uterine transplantation — Transplantation of the uterus from live donor and IVF treatment.

SUMMARY:
Uterus transplantation, as a possible future treatment for uterine factor infertility, has been developed in animal species during the last decade.

The study protocol includes transplantation of the uterus from a live donor (mother, relative, friend) into women with absolute uterine factor infertility (lack of uterus from birth or due to life saving hysterectomy).The recipient will be treated by standard immunosuppression and transfer of embryos (acquired by IVF before surgery) will be attempted when at least 12 months have passed from transplantation. Approval for a case series including up to 10 patients has been acquired.

DETAILED DESCRIPTION:
The study is ongoing, with inclusion of 9 patients.

ELIGIBILITY:
Inclusion Criteria:

* less than 39 years
* good general health

Exclusion Criteria:

* poor ovarian resaerve or older than 39 years
* systemic or psychiatric disease

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
surviving transplants (12 months) | up to 3 years after transplantation

SECONDARY OUTCOMES:
pregnancy rate | up to 3 years after transplantation

OTHER OUTCOMES:
live birth rate | up to 4 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mats Brännström, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Mats Brännström, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Scientific publications

REFERENCES:
- [Background] Jarvholm S, Kattstrom A, Kvarnstrom N, Dahm-Kahler P, Brannstrom M. Long-term health-related quality-of-life and psychosocial outcomes after uterus transplantation: a 5-year follow-up of donors and recipients. Hum Reprod. 2024 Feb 1;39(2):374-381. doi: 10.1093/humrep/dead245. PMID 37995381
- [Background] Jarvholm S, Bokstrom H, Enskog A, Hammarling C, Dahm-Kahler P, Brannstrom M. Striving for motherhood after uterus transplantation: a qualitative study concerning pregnancy attempts, and the first years of parenthood after transplantation. Hum Reprod. 2022 Jan 28;37(2):274-283. doi: 10.1093/humrep/deab260. PMID 34865019
- [Background] Jarvholm S, Dahm-Kahler P, Kvarnstrom N, Brannstrom M. Psychosocial outcomes of uterine transplant recipients and partners up to 3 years after transplantation: results from the Swedish trial. Fertil Steril. 2020 Aug;114(2):407-415. doi: 10.1016/j.fertnstert.2020.03.043. Epub 2020 Jul 22. PMID 32709381
- [Background] Jarvholm S, Enskog A, Hammarling C, Dahm-Kahler P, Brannstrom M. Uterus transplantation: joys and frustrations of becoming a 'complete' woman-a qualitative study regarding self-image in the 5-year period after transplantation. Hum Reprod. 2020 Aug 1;35(8):1855-1863. doi: 10.1093/humrep/deaa143. PMID 32619006
- [Background] Jarvholm S, Kvarnstrom N, Dahm-Kahler P, Brannstrom M. Donors' health-related quality-of-life and psychosocial outcomes 3 years after uterus donation for transplantation. Hum Reprod. 2019 Jul 8;34(7):1270-1277. doi: 10.1093/humrep/dez087. PMID 31241745
- [Background] Broecker V, Brannstrom M, Bosmuller H, Sticova E, Maluskova J, Chiesa-Vottero A, Molne J. Reproducibility of Rejection Grading in Uterus Transplantation: A Multicenter Study. Transplant Direct. 2023 Sep 20;9(10):e1535. doi: 10.1097/TXD.0000000000001535. eCollection 2023 Oct. PMID 37745947
- [Background] Karlsson CC, Dahm-Kahler P, Kvarnstrom N, Molne J, Broecker V, Brannstrom M. Hysterectomy after uterus transplantation and detailed analyses of graft failures. Acta Obstet Gynecol Scand. 2022 Mar;101(3):355-363. doi: 10.1111/aogs.14304. Epub 2021 Dec 14. PMID 34907538
- [Background] Broecker V, Brannstrom M, Ekberg J, Dahm-Kahler P, Molne J. Uterus transplantation: Histological findings in explants at elective hysterectomy. Am J Transplant. 2021 Feb;21(2):798-808. doi: 10.1111/ajt.16213. Epub 2020 Aug 11. PMID 32659865
- [Background] Molne J, Broecker V, Ekberg J, Nilsson O, Dahm-Kahler P, Brannstrom M. Monitoring of Human Uterus Transplantation With Cervical Biopsies: A Provisional Scoring System for Rejection. Am J Transplant. 2017 Jun;17(6):1628-1636. doi: 10.1111/ajt.14135. Epub 2017 Jan 3. PMID 27868389
- [Result] Brannstrom M, Bokstrom H, Dahm-Kahler P, Diaz-Garcia C, Ekberg J, Enskog A, Hagberg H, Johannesson L, Kvarnstrom N, Molne J, Olausson M, Olofsson JI, Rodriguez-Wallberg K. One uterus bridging three generations: first live birth after mother-to-daughter uterus transplantation. Fertil Steril. 2016 Aug;106(2):261-6. doi: 10.1016/j.fertnstert.2016.04.001. Epub 2016 Apr 25. PMID 27125227
- [Result] Johannesson L, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Diaz-Garcia C, Olausson M, Brannstrom M. Uterus transplantation trial: 1-year outcome. Fertil Steril. 2015 Jan;103(1):199-204. doi: 10.1016/j.fertnstert.2014.09.024. Epub 2014 Oct 22. PMID 25439846
- [Result] Brannstrom M, Johannesson L, Bokstrom H, Kvarnstrom N, Molne J, Dahm-Kahler P, Enskog A, Milenkovic M, Ekberg J, Diaz-Garcia C, Gabel M, Hanafy A, Hagberg H, Olausson M, Nilsson L. Livebirth after uterus transplantation. Lancet. 2015 Feb 14;385(9968):607-616. doi: 10.1016/S0140-6736(14)61728-1. Epub 2014 Oct 6. PMID 25301505
- [Result] Brannstrom M, Johannesson L, Dahm-Kahler P, Enskog A, Molne J, Kvarnstrom N, Diaz-Garcia C, Hanafy A, Lundmark C, Marcickiewicz J, Gabel M, Groth K, Akouri R, Eklind S, Holgersson J, Tzakis A, Olausson M. First clinical uterus transplantation trial: a six-month report. Fertil Steril. 2014 May;101(5):1228-36. doi: 10.1016/j.fertnstert.2014.02.024. Epub 2014 Feb 27. PMID 24582522
- [Result] Jarvholm S, Johannesson L, Clarke A, Brannstrom M. Uterus transplantation trial: Psychological evaluation of recipients and partners during the post-transplantation year. Fertil Steril. 2015 Oct;104(4):1010-1015. doi: 10.1016/j.fertnstert.2015.06.038. Epub 2015 Jul 28. PMID 26231464
- [Result] Jarvholm S, Johannesson L, Brannstrom M. Psychological aspects in pre-transplantation assessments of patients prior to entering the first uterus transplantation trial. Acta Obstet Gynecol Scand. 2015 Oct;94(10):1035-8. doi: 10.1111/aogs.12696. Epub 2015 Jun 30. PMID 26073658
- [Result] Brannstrom M, Dahm-Kahler P, Kvarnstrom N, Enskog A, Olofsson JI, Olausson M, Molne J, Akouri R, Jarvholm S, Nilsson L, Stigson L, Hagberg H, Bokstrom H. Reproductive, obstetric, and long-term health outcome after uterus transplantation: results of the first clinical trial. Fertil Steril. 2022 Sep;118(3):576-585. doi: 10.1016/j.fertnstert.2022.05.017. Epub 2022 Jun 11. PMID 35697530
- [Derived] Wentz E, Hagberg B, Hagberg H, Bokstrom H, Brannstrom M. Uterus transplantation; first data on neurologic, neuropsychiatric, and physical examination follow-up of children up to 6 years of age. Hum Reprod. 2025 Dec 1;40(12):2419-2429. doi: 10.1093/humrep/deaf178. PMID 40971624
- [Derived] Brannstrom M, Ekberg J, Sandman L, Davidson T. The costs per live birth after uterus transplantation: results of the Swedish live donor trial. Hum Reprod. 2025 Feb 1;40(2):310-318. doi: 10.1093/humrep/deae272. PMID 39675045
- [Derived] Carbonnel M, Petit M, Tarantino N, Morin V, Corneau A, Tourne M, Gueguan J, Molne J, Akouri R, Broecker V, Vinit A, Racowsky C, Brannstrom M, Ayoubi JM, Vieillard V. Analysis of Immunological Biomarkers Associated With Rejection After Uterus Transplantation in Human. Transplantation. 2025 Feb 1;109(2):e119-e133. doi: 10.1097/TP.0000000000005126. Epub 2024 Jul 18. PMID 39020469
- [Derived] Davidson T, Ekberg J, Sandman L, Brannstrom M. The costs of human uterus transplantation: a study based on the nine cases of the initial Swedish live donor trial. Hum Reprod. 2021 Jan 25;36(2):358-366. doi: 10.1093/humrep/deaa301. PMID 33247912